CLINICAL TRIAL: NCT03589235
Title: Evaluation of the Usage of Platelet-Rich Fibrin Dressing in the Management of Free Gingival Graft and Donor Site Palatal Wound
Brief Title: Platelet-Rich Fibrin Dressing in the Management of Free Gingival Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Perio-02-2018
Record Dates: First submitted 2018-07-02; First posted 2018-07-17 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Gingival Recession
Keywords: autografts; gingival recession; free gingival graft; Attached gingival width; Platelet-Rich Fibrin dressing
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Platelet-Rich Fibrin dressing (Experimental): A Platelet-Rich Fibrin dressing (PRF) will be used in both donor and receiving sites after a free gingival graft.
  Interventions: Procedure: A free gingival graft; Device: A Platelet-Rich Fibrin dressing
- A non-eugenol-based dressing (Experimental): A non-eugenol-based dressing (Coe-Pak™) will be used in both donor and receiving sites after a free gingival graft.
  Interventions: Procedure: A free gingival graft; Device: A non-eugenol-based dressing

INTERVENTIONS:
Procedure: A free gingival graft — A free gingival graft will be used for the treatment of gingival recession
Device: A Platelet-Rich Fibrin dressing — A Platelet-Rich Fibrin dressing (PRF) will be applied in both donor and receiving sites after the free gingival graft.
  Arms: A Platelet-Rich Fibrin dressing
Device: A non-eugenol-based dressing — A non-eugenol-based dressing (Coe-Pak™) will be applied in both donor and receiving sites after the free gingival graft.
  Arms: A non-eugenol-based dressing

SUMMARY:
Evaluation of two dressing materials; a Platelet-Rich Fibrin (PRF) dressing and a non-eugenol-based (Coe-Pak™) dressing in the management of free gingival graft and donor site palatal wound.

DETAILED DESCRIPTION:
Evaluation of the usage of platelet-rich fibrin dressing in the management of free gingival graft and donor site palatal wound by evaluation of pain score, healing tissue in both donor and receiving sites, coverage of gingival recession, and the gain of attached gingiva.

A total of 20 subjects will be invited to participate in this study from the patients seeking treatment at the Department of Periodontology, Faculty of Dentistry, Damascus University.

The study has been approved by the investigator's local Review Board. Subjects will be recruited according to specific inclusion criteria. After completion of medical and dental history questionnaires, patients will sign a consent form after being advised about the nature of the study.

Patients will be allocated into two groups (10 patients each). A Platelet-Rich Fibrin (PRF) dressing will be used in both donor and receiving sites in the test group, while a non-eugenol-based (Coe-Pak™) dressing will be used in both donor and receiving sites in the control group .

Donor site working time, bleeding (BLE), colour match (CM), pain and re-epithelization (EP) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Syrian descent.
* Systemically healthy.
* Attached gingival width ≤ 2 mm.
* Presence of type II (Miller Classification) of gingival recession.

Exclusion Criteria:

* Smoking.
* Pregnancy or lactating.
* Presence of any systematic diseases can affect the periodontal surgery.
* Subjects with significant moderate to severe periodontal disease.
* Patients under orthodontic treatment
* Presence of restorative materials (e.g. crown)
* Subjects have failed to maintain good plaque control.
* Subjects having previous surgical treatment for covering the recession in the chosen area.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
The pain score using the visual analogue scale (VAS) | The Pain score will be evaluated twice. At T1 (after 2 days of surgery) and T2 (after 7 days of surgery).
  This variable is going to be measured by an visual analogue scale (VAS). The VAS pain scores ranges between 0 to10. (0: no pain, 1: minimal pain, 10: severe pain).

SECONDARY OUTCOMES:
Healing index for free gingival graft | The healing index will be evaluated twice. At T1 (after one week of surgery) and T2 (after one month of surgery)..
  The healing index for free gingival graft is an ordinal score: very poor, poor, good, very good and excellent.
The complete re-epithelialization of the palatal wound | The measurements will be performed at T1 (after 1 week measurement), T2 (after 2 weeks measurement), T3 (after 3 weeks measurement), and T4 (after 4 weeks measurement).
  This variable is going to be measured using the peroxide test. Scores are yes or no for showing bubbles.
Changes in gingival recession | The measurement will be performed at T0 (baseline measurement) and at T1 (at three months exactly post-operatively measurement).
  Miller Class II of Gingival recession is measured from the cemento-enamel junction to the gingival margin of the recessed tissues.
Match color of the palatal wound | The measurement will be performed at T1 (after 1 week measurement) and T2 (after 1 month measurement).
  VAS scores (between 0 and 10. 0: no CM, 10: excellent CM) in comparison with adjacent and contralateral palatal mucosa.
Attached gingival width | The measurement will be performed at T0 (baseline measurement) and at T1 (after 3 months measurement).
  Measured from the Mucogingival junction to the gingival Groove.
Plaque index | The measurement will be performed at T0 (baseline measurement) and at T1 (at three months exactly post-operatively measurement).
  Score: none, simple, middle, severe.
Gingival Index | The measurement will be performed at T0 (baseline measurement) and at T1 (at three months exactly post-operatively measurement).
  Score: none, simple, middle. Severe.
Bleeding on probing Index | The measurement will be performed at T0 (baseline measurement) and at T1 (at three months exactly post-operatively measurement).
  Score: bleeding, none bleeding.
Pocket Probing Depth | The measurement will be performed at T0 (baseline measurement) and at T1 (at three months exactly post-operatively measurement).
  Score: normal, simple, middle, severe.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Abou Sulaiman, PhD., Study Director — Department of Orthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No
The Individual participant data will be only available for the researchers in the department of Periodontics, Damascus University

REFERENCES:
- [Result] Bansal M, Kumar A, Puri K, Khatri M, Gupta G, Vij H. Clinical and Histologic Evaluation of Platelet-Rich Fibrin Accelerated Epithelization of Gingival Wound. J Cutan Aesthet Surg. 2016 Jul-Sep;9(3):196-200. doi: 10.4103/0974-2077.191647. PMID 27761092
- [Result] Femminella B, Iaconi MC, Di Tullio M, Romano L, Sinjari B, D'Arcangelo C, De Ninis P, Paolantonio M. Clinical Comparison of Platelet-Rich Fibrin and a Gelatin Sponge in the Management of Palatal Wounds After Epithelialized Free Gingival Graft Harvest: A Randomized Clinical Trial. J Periodontol. 2016 Feb;87(2):103-13. doi: 10.1902/jop.2015.150198. Epub 2015 Aug 27. PMID 26313017
- [Result] Keceli HG, Aylikci BU, Koseoglu S, Dolgun A. Evaluation of palatal donor site haemostasis and wound healing after free gingival graft surgery. J Clin Periodontol. 2015 Jun;42(6):582-9. doi: 10.1111/jcpe.12404. Epub 2015 May 19. PMID 25892528
- [Result] Keskiner I, Lutfioglu M, Aydogdu A, Saygun NI, Serdar MA. Effect of Photobiomodulation on Transforming Growth Factor-beta1, Platelet-Derived Growth Factor-BB, and Interleukin-8 Release in Palatal Wounds After Free Gingival Graft Harvesting: A Randomized Clinical Study. Photomed Laser Surg. 2016 Jun;34(6):263-71. doi: 10.1089/pho.2016.4094. Epub 2016 Apr 18. PMID 27088277
- [Result] Ustaoglu G, Ercan E, Tunali M. The role of titanium-prepared platelet-rich fibrin in palatal mucosal wound healing and histoconduction. Acta Odontol Scand. 2016 Oct;74(7):558-564. doi: 10.1080/00016357.2016.1219045. Epub 2016 Aug 19. PMID 27538770
- [Result] Shanmugam M, Kumar TS, Arun KV, Arun R, Karthik SJ. Clinical and histological evaluation of two dressing materials in the healing of palatal wounds. J Indian Soc Periodontol. 2010 Oct;14(4):241-4. doi: 10.4103/0972-124X.76929. PMID 21731250